CLINICAL TRIAL: NCT05883189
Title: Establish the Reference Range of Antiphospholipid Antibody in Healthy Preganany Women: The Prospective Studies for Antiphospholipid Syndrome Related Pregancy Loss
Brief Title: Establish the Referenc Range of Antiphospholipid Antibody in Healthy Preganany Women
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, chenhui79, Chief Physician, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Other Study IDs: SYSKY-2022-412-01
Record Dates: First submitted 2023-05-20; First posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Focus Health Pregancy Women

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (3):
- Group1: non-pregancy health women.
  Interventions: Diagnostic Test: Draw blood
- Group 2:Pregancy health women.
  Interventions: Diagnostic Test: Draw blood
- Group 3: Diagnosed Antiphospholipid syndrome patients
  Interventions: Diagnostic Test: Draw blood

INTERVENTIONS:
Diagnostic Test: Draw blood — Draw blood from human body and make into serum to test

SUMMARY:
The study is aim to establish 95th and 99th percentile for healthy pregancy women for antiphospholipid antibodies(aPLs), such as aCL IgG/M/A, B2GP1 IgG/M/A, aPS/PT IgG/M. The outcome of the study is expected to aid Antiphospholipid syndrome patients diagnosis and managment. We also include some obstetirc Antiphospholipid syndrome(APS) patients to analysis the correlation between antiphospholipid antibodies and pregancy outcome, also want to know the prevalenc of aPLs, which can be guide for clinical application for APS diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

* 120 non-pregnant healthy women, Age 18-45, with at least 1 successful pregnancy , no history of adverse pregnancy outcome, no abortion, still birth, premature delivery, preeclampsia
* 120 pregnant women, Age 18-45, follow through the pregnancy and successful delivery without any adverse pregnancy outcome during the pregnancy process, no abortion, still birth, premature delivery, preeclampsia, no drug treatment
* 60 APS pregnant patients diagnosed by clinical department

Exclusion Criteria:

1. Thrombosis history
2. Rheumatic immune disease
3. Use oral contraception or biological inhibitors
4. History of abortion, adverse pregnancy outcome, common high blood pressure, diabetes

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 1. Non-pregnant healthy women, Age 18-45;
  2. Pregnant women, Age 18-45, follow through the pregnancy and successful delivery
  3. APS pregnant patients diagnosed by clinical department
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-05-20 (Estimated); Primary Completion 2023-10-07 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
95th and 99th pencentile data of pregancy and non-pregancy women | Oct. 2023
  95th and 99th pencentile data of pregancy and non-pregancy women, and the prevalence of aPLs

IPD SHARING:
Plan to Share IPD: Undecided